CLINICAL TRIAL: NCT07189299
Title: Role of the Serotonin 2A Receptor in Women With Premenstrual Disorders: a Randomized, Double-blind, Placebo-controlled Study (L4Her-Study)
Brief Title: Microdosing LSD in Women With Premenstrual Disorders
Acronym: L4Her
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Friederike Holze (Other)
Responsible Party: Sponsor-Investigator, Friederike Holze, Head of Clinical Research, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BASEC 2025-00745
Record Dates: First submitted 2025-08-22; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: PMS; PMDD
Keywords: Hallucinogens; Serotonin Agents; LSD; Premenstrual disorders; Premenstrual syndrome; Psychotropic drugs; Microdose; Serotonin system; Psychedelics
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, placebo-controlled, parallel design with 3 intervention arms. Participants will be allocated in a 1:1:1 ratio to one arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 μg LSD every day during the acute symptom phase (Experimental): Participants receive 10 μg LSD daily, starting at symptom onset (or latest 7 days after ovulation) until day 3 of the following cycle for 3 menstrual cycles
  Interventions: Drug: LSD 10 μg every Day
- 10 μg LSD every second day during acute symptom phase (Experimental): 10 μg LSD every second day during acute symptom phase starting at symptom onset (or 7 days after ovulation) until day 3 of the following cycle for 3 menstrual cycles
  Interventions: Drug: LSD 10 μg every other day
- Placebo Control (Placebo Comparator): The subjects in the control arm will receive oral placebo over 3 cycles during the luteal phase, starting at symptom onset (or latest 7 days after ovulation) until day 3 of the following cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LSD 10 μg every Day — Participants will receive 10 μg LSD every day during the luteal phase
  Arms: 10 μg LSD every day during the acute symptom phase
Drug: LSD 10 μg every other day — Participants receive 10μg LSD every second day during the luteal phase
  Arms: 10 μg LSD every second day during acute symptom phase
Drug: Placebo — Participants receive inactive placebo during the luteal phase
  Arms: Placebo Control

SUMMARY:
The investigators aim to investigate the role of the serotonin 2A receptor in women with premenstrual disorders. This study uses a double-blind, randomized, controlled design with 3 arms: Intervention 1: 10 micg LSD for ~10 days during the late luteal phase (for 3 cycles) Intervention 2: 10 micg LSD every other day for ~10 days during the late luteal phase (for 3 cycles) Control intervention: Placebo for ~10 days during the late luteal phase (for 3 cycles) Each participant will be treated in only one arm. The study employs a parallel design with three treatment arms and consists of a two-cycle observational phase followed by a three-cycle treatment phase.

DETAILED DESCRIPTION:
Premenstrual disorders (premenstrual syndrome (PMS) and Premenstrual Dysphoric Disorder (PMDD)) affect many women (20 - 30% for PMS and 1.2 - 6.4% for PMDD) and are associated with affective symptoms, pain, mood impairment, insomnia, loss of well-being, and productivity making it complex disorders with combined mood, physical, and cognitive symptoms.

The serotonin 2A receptor has been shown to be potentially involved in the pathophysiology of premenstrual disorders, however the mechanism remains to be investigated. Anecdotal evidence suggests that low doses of psychedelics like LSD or psilocybin, taken during the luteal phase, may help alleviate symptoms. However, this approach lacks scientific validation and requires further research. We therefore seek to investigate if repeated and targeted administration of low doses of the serotonin 2A receptor agonist LSD modulates the symptom burden in premenstrual disorders.

The study employs a parallel design with three treatment arms and consists of a two-cycle observational phase followed by a three-cycle treatment phase. Timepoints below are based on a 28-day menstrual cycle, but will be adapted based on individual menstrual cycle durations.

ELIGIBILITY:
Inclusion crtieria:

* Between 18-45 years.
* Are menstruating and have cycles with a duration between 21 - 35 days.
* Meet DSM-V criteria for PMDD or criteria for severe PMS with daily ratings over 2 cycles to confirm luteal symptoms.

  1. For PMDD, participants must have a minimal average luteal phase score of mild (≥3 on a 6-point scale) for at least 5 Symptoms on the DRSP including 1 mood symptom during the 5 most symptomatic of the final 7 luteal phase days and the first 2 days of menses onset, and the average follicular phase score must not be >2 on these same items.
  2. For severe PMS, participants must have a minimal average luteal phase score of mild (≥3 on a 6-point scale) for at least 4 Symptoms on the DRSP including 1 mood symptom, during the 5 most symptomatic of the final 7 luteal phase days and the first 2 days of menses onset, and the average follicular phase core must not be >2 on these same items.
* Have reported PMDD/PMS symptoms for the majority of menstrual cycles (>9 of 12) during the year prior to screening.
* Sufficient understanding of the German language
* Sufficient understanding of the study procedures and risks associated with the study.
* Participants must be willing to adhere to the study procedures and sign the consent form.
* Willing not to drive or operate heavy machinery during the acute treatment phases of the study.
* Willing to refrain from more than 7 standard alcoholic drinks a week, more than 10 cigarettes a day, and any illicit substances.
* Willing to use effective contraceptive measures throughout study participation.

Exclusion Criteria:

* Known hypersensitivity to LSD
* Current treatment for PMS/PMDD
* Use of an oral hormonal contraceptive < 6 months.
* Past or present bipolar or psychotic disorder, including depressive disorder with psychotic features.
* First degree relative with a psychotic disorder.
* Significant prodromal psychotic symptoms (Prodromal Questionnaire-16 symptoms ≥ 6).
* Borderline personality disorder.
* Current post-traumatic stress disorder.
* Pregnant or breastfeeding
* Planned pregnancy.
* Current or recent history of significant suicide ideation or suicide behavior within the past 6 months.
* Current substance use disorder (< 12 months) other than tobacco smoking.
* Other illness that excludes repeated LSD administration or requires interfering medication.
* Participation in another clinical trial (currently or within the last 30 days)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in premenstrual symptom burden | Daily over the 5 cycle study course (average cycle duration is 28 days)
  Premenstrual symptom burden measured with the Daily Record of Severity of Problems (DRSP) total score as the mean of the 5 highest symptomatic days of the 7 days before menstruation onset as mean change from baseline (the two monitored cycles before treatment start) of symptoms over all three treatment periods compared with the other study arms.

SECONDARY OUTCOMES:
Montgomery-Asberg-Depression-Rating Scale (MARDS) | Ratings will be performed on day 3 of each menstural cycle, over the whole study period of 5 menstrual cycles, to retrospectively rate depressive symptoms during the premenstrual phase (based on an average cycle duration of 28 days)
  The Montgomery-Asberg-Depression Rating Scale (MADRS) is a ten-item questionnaire widely used to measure severity of depressive symptoms.
Hamilton Anxiety Rating Scale (HAM-A) | Ratings will be performed on day 3 of each menstural cycle , over the whole study period of 5 menstrual cycles to retrospectively rate anxiety symptoms during the premenstrual phase ((based on an average cycle duration of 28 days).
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-rated scale developed to measure the severity of anxiety symptoms.
State-trait anxiety inventory (STAI) | The STAI will be repeatedly assessed 3 times per cycle (twice during the late luteal phase (cycle day 20 and 26 based on a 28-day cycle) and on day 3 after start of mensturation) over the whole study period of 5 menstrual cycles.
  The State-trait anxiety inventory (STAI) is a widely used self-report instrument for assessing anxiety in adults. It includes separate measures of state and trait anxiety.
Beck Depression Inventory (BDI) | The BDI will be repeatedly assessed 3 times per cycle (twice during the late luteal phase (cycle day 20 and 26 based on a 28-day cycle) and on day 3 after start of mensturation) over the whole study period of 5 menstrual cycles.
  The BDI consists of 21 questions developed to measure depression severity. In contrast to the MADRS, the BDI is a self-rating instrument.
Quality of Life (WHOQOL-bref) | The WHOQOL-bref will be repeatedly assessed 3 times per cycle (twice during the late luteal phase (cycle day 20 and 26 based on a 28-day cycle) and on day 3 after start of me, additionally it will be assessed at screening and once during the luteal phase
  The WHOQOL-bref (World Health Organization Quality of life scale) is one of the most commonly used self-rating instruments for the assessment of the quality of life. The scale includes 26 items and four domain scores can be derived (physical, psychological, social relationships, and environmental).
Menstrual pain | Menstrual pain will be assessed on menstruation days over 5 menstrual cycles (average cycle duration is 28 days).
  Menstrual pain will be assessed via 3 main questions. 1.) Did you experience any menstruation-related pain today? (VAS 0-100) 2.) Did you do anything for pain relief? (YES / NO). If "YES" 3a.) Did you take any medication? If yes, what, how much and how often? 3b.) Did you conduct any non-drug treatment? If yes, what, how much and how often? 3c.) Other? (free answer).
Quality of Sleep | Participants are asked to rate their sleep quality daily over 5 menstrual cycles (average cycle duration is 28 days).
  Rating consists of 5 questions. 1. How did you sleep? (bidirectional VAS from -50 very bad to 50 very good). 2. How fast did you fall asleep (bidirectional VAS from -50 very fast to 50 not at all) 3. Did you wake-up during the night? (YES/NO, if YES, how many times?) 4. Do you feel refreshed? (bidirectional VAS from -50 not at all to 50 very much) 5. Did you have a hard time waking-up this morning? (bidirectional VAS from -50 not at all to 50 very much).
Daily mood (AMRS) | The AMRS will be administered daily over 5 menstrual cycles (average cycle duration is 28 days).
  The Adjective Mood Rating Scale (AMRS or EWL60S) is a 60-item Likert scale that allows repeated assessment of mood.
Female Sexual Function Index (FSFI) | The outcome will be on day 3 of each menstural cycle to retrospectively rate sexual function during the premenstrual phase over 5 menstrual cycles (average cycle duration is 28 days).
  The FSFI is a comprehensive, validated tool designed to assess key dimensions of sexual function in women.
Concomitant Medication | Complete concomitant medication including on-demand medication during bleeding days (dysmenorrhea) will be assessed at screening and rescreening. The exact intake will be recorded daily over 5 menstrual cycles (average cycle duration is 28 days).
  Intake of pain medication during acute treatment phases and menstruation
Subjective effects questionnaire (Visual Analog Scales, VAS) | Will be assessed during the first drug administration in cycle 3, latest 7 days after ovulation (average cycle duration is 28 days). Scales will be administered at 0, 0.5, 1, 2, 3, 4, 5, and 6 hours after substance administration.
  VAS will be repeatedly used during the first drug sessions to assess subjective effects. The following VAS will be used: "any drug effect", "good drug effect", "bad drug effect", "liking", "high", "anxiety". The maximal ratings (Emax, 0-100) and area under the effect curve (AUEC) values will be defined for each VAS item and Emax and AUEC values will be compared between treatments using ANOVAs.
5-Dimensions of Altered States of Consciousness (5D-ASC) | Only once 6 hours after drug administration on the first in-house drug application (cycle 3, latest 7 days after ovulation, average cycle duration is 28 days)
  The 5 Dimensions of Altered States of Consciousness (5D-ASC) Scale is a questionnaire containing visual analog scales for 94 items to restrospectively assess peak alterations in state of consciousness.
Mystical Effects Questionnaire (MEQ) | Only once 6 hours after drug administration on the first in-house drug application (cycle 3, latest 7 days after ovulation, average cycle duration is 28 days)
List of complaints (LC) | Twice during the first in-house drug application (cycle 3, latest 7 days after ovulation, average cycle duration is 28 days) baseline (before drug administration) and 6 hours after drug administration.
  The list of complaints (LC) consists consists of a 40-items list to assess physiological complaints throughout the study.
Changes in cognition | Once during the luteal phase of an unmedicated cycle (cycle day 26 based on a 28-day cycle), once during the luteal phase of a medicated cycle (cycle day 26 based on a 28-day cycle), and once during the follicular phase of a medicated cycle.
  Cognition will be assessed using CANTAB tasks.
Blood pressure | Will be assessed during the first drug administration in cycle 3, latest 7 days after ovulation -0.5, 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5 and 6 hours after substance administration (average cycle duration is 28 days).
  Systolic and diastolic blood pressure will be repeatedly measured during the first drug administration.
Heart rate | Will be assessed during the first drug administration in cycle 3, latest 7 days after ovulation -0.5, 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5 and 6 hours after substance administration (average cycle duration is 28 days).
Expectancy as mediator for treatment effects | Baseline
  To measure expectancy, we will use a modified 2-item version of the Credibility / Expectancy Questionnaire (CEQ).
Personality traits as mediator for treatment effects (NEO-FFI) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The NEO Five Factor Inventory (NEO-FFI) is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness.
Personality traits as mediator for treatment effects (FPI-R) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Freiburger Personality Inventory (FPI-R) version comprises 138 items and covers 12 dimensions of personality.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No